CLINICAL TRIAL: NCT05889442
Title: Effect of Levcromakalim in Individuals With Migraine Pretreated With Erenumab: A Randomized Double-Blind Placebo-Controlled Two-Way Crossover Trial
Brief Title: Effect of Levcromakalim in Individuals With Migraine Pretreated With Erenumab
Acronym: COLLIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Messoud Ashina, MD, Professor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-22031695
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Cromakalim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Experimental)
  Interventions: Drug: Levcromakalim
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levcromakalim — Continuous intravenous infusion of 20 mL levcromakalim (0.05 mg/min (50 μg/ mL) over 20 minutes
  Arms: Levcromakalim
Other: Placebo — Continuous intravenous infusion of 20 mL isotonic saline over 20 minutes
  Arms: Placebo

SUMMARY:
An outstanding scientific question, that merits further investigation, is whether dilation of intracranial arteries is implicated in the pathogenesis of cephalic pain in migraine. Here, we hypothesize that experimentally-induced dilation of intracranial arteries using intravenous infusion of levcromakalim (a potent vasodilator) induces cephalic pain with migraine-like features in people with migraine, who prior to the infusion are administered erenumab (anti-calcitonin gene-related peptide (CGRP) receptor monoclonal antibody).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study-specific activities/procedures.
* Age ≥18 years upon entry into screening.
* History of migraine without aura for ≥12 months with a frequency of 1-5 migraine attacks per month before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018), based on medical records and/or patient self-report.

Exclusion Criteria:

* History of any primary headache disorder other than migraine without aura, or tension-type headache with a frequency of ≥5 headache days per month before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018), based on medical records and/or patient self-report.
* History of any secondary headache disorder before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018) based on medical records and/or patient self-report.
* Intake of prophylactic migraine medication within ≤30 days or 5 plasma half-lives (whichever is longer) prior to screening.
* Prior intake of therapies targeting the CGRP signaling pathway, including anti-CGRP ligand monoclonal antibodies, anti-CGRP receptor monoclonal antibodies, and small molecule CGRP receptor antagonists.
* The participant is at risk of self-harm or harm to others as evidenced by past suicidal behavior.
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator will pose a risk to participant safety or interfere with the study evaluation, procedures or completion.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a urine pregnancy test.
* Female participants who are pregnant or breastfeeding or plan to become pregnant or breastfeed during participation in the study.
* Evidence of current pregnancy or breastfeeding per participant self-report or medical records.
* Participants likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participants' and investigator's knowledge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence of migraine attack | 12 hours
  Difference in incidence of migraine attack (0 to 12 hours) between levcromakalim and placebo.
  A migraine attack is defined as an attack fulfilling either (i) or (ii):
  (i)* Headache fulfilling criteria C and D for migraine without aura according to the International Headache Society criteria:
  C. Headache has at least two of the following characteristics:
  unilateral location pulsating quality moderate or severe pain intensity (moderate to severe pain intensity is considered ≥4 on verbal rating scale) aggravation by cough (in-hospital phase) or causing avoidance of routine physical activity (out-hospital phase)
  D. During headache at least one of the following:
  nausea and/or vomiting photophobia and phonophobia (ii) Headache described as mimicking the patient's usual migraine attack and treated with acute migraine medication (rescue medication).

SECONDARY OUTCOMES:
Incidence of headache | 12 hours
  Difference in incidence of headache (0 to 12 hours) between levcromakalim and placebo.
  Incidence of headache is defined as headache intensity ≥1 as measured by a numerical rating scale (NRS) from 0 to 10. It is a verbally declared scale from 0 to 10, where 0 is no pain; 10 is the worst pain imaginable.
Intensity of headache | 12 hours
  Difference in area under the curve (AUC) for headache intensity scores (0 to 12 hours) between levcromakalim and placebo.
  Headache intensity scores are measured by a numerical rating scale (NRS). It is a verbally declared scale from 0 to 10, where 0 is no pain; 10 is the worst pain imaginable.
Diameter of superficial temporal artery | 1 hour
  Diameter (mm) of superficial temporal artery is measured as a continuous outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Denmark

REFERENCES:
- [Derived] Raffaelli B, Do TP, Chaudhry BA, Amin FM, Ashina H, Snellman J, Maio-Twofoot T, Ashina M. Activation of ATP-sensitive potassium channels triggers migraine attacks independent of calcitonin gene-related peptide receptors: a randomized placebo-controlled trial. Cephalalgia. 2024 Jan;44(1):3331024231222916. doi: 10.1177/03331024231222916. PMID 38181724